CLINICAL TRIAL: NCT03744455
Title: Influence of Resident's Degree of Formation on the Quality of Care Delivered to the Patients.
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, FAHA, Head of Department, Astes
Other Study IDs: PQR
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- End of training: Anesthesia residents at the end of their training who will realize axillary plexus. The satisfaction of the patient will be registered.
  Interventions: Biological: Axillary Plexus
- Begin of training: Anesthesia residents at the begin of their training who will realize axillary plexus. The satisfaction of the patient will be registered.
  Interventions: Biological: Axillary Plexus

INTERVENTIONS:
Biological: Axillary Plexus — Axillary plexus anesthesia technique for hand surgery

SUMMARY:
The aim of this study is to evaluation the influence of the resident in anesthesiology's degree of formation on the quality of care delivered to the patient.

DETAILED DESCRIPTION:
The aim of this study is to evaluation the influence of the resident in anesthesiology's degree of formation on the quality of care delivered to the patient.

To perform it, the investigators will enrolled all of the patients scheduled for an axillary plexus anesthesia technique in the Clinique Saint-Luc of Bouge in September 2018 (end of formation for the residents in anesthesia) and compare the patient's degree of satisfaction with the patients scheduled for the same kind of anesthesia on October and November 2018 (begin of formation for the residents in anesthesia).

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for hand surgery under axillary plexus

Exclusion Criteria:

* Patient's refusal

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for hand surgery under axillary plexus in the Clinique Saint-Luc of Bouge (Namur, Belgium)
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction (Likert's scale) | 1 day
  Patient satisfaction after the completion of axillary plexus (satisfaction will be studied with a Lickert's scale). This scale will examine the patient's satisfaction in a scale ranging from 0 (worse satisfaction) to 5 (best satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deflandre, MD, PhD, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc Bouge, Namur, Belgium